CLINICAL TRIAL: NCT00388427
Title: Phase I Study of Cetuximab Plus Dasatinib (BMS-354825) in Advanced Solid Malignancies
Brief Title: Safety Study Of Cetuximab Plus Dasatinib (BMS-354825) in Treating Advanced Solid Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Edward Chu, MD, Principal Investigator, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-038; CA180049 (Other: BMS)
Record Dates: First submitted 2006-10-13; First posted 2006-10-16 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2014-01

CONDITIONS: Malignant Solid Tumour
Keywords: advanced cancer; solid tumor; solid malignancies; phase I
MeSH Terms: interventions — Dasatinib; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Advanced Solid Malignancies (Other)
  Interventions: Drug: Dasatinib (BMS-354825); Drug: Cetuximab (Erbitux, C225)

INTERVENTIONS:
Drug: Dasatinib (BMS-354825) — 100 mg, 150 mg, or 200 mg per dose escalation schedule; continuous oral dosing on Days 1-21 of each 21-day cycle until progression or unacceptable toxicity develops.
Drug: Cetuximab (Erbitux, C225) — Loading dose of IV 400 mg/m^2 on Day 1 of Cycle 1; IV 250 mg/m^2 weekly thereafter each 21-day cycle until progression or unacceptable toxicity develops.

SUMMARY:
This is an open-label, safety study of cetuximab and differing dose levels of dasatinib in adult patients with advanced solid malignancies. Cetuximab will be administered as an intravenous infusion weekly. Dasatinib will be taken orally, once a day, on a continuous schedule at differing dose levels. The primary objective of this study is to determine the toxicities and the maximum tolerated doses of dasatinib when combined with cetuximab for the treatment of advanced solid tumors.

DETAILED DESCRIPTION:
This is an open-label, phase I study of cetuximab and differing dose levels of dasatinib in adult patients with advanced solid malignancies. Cetuximab will be administered as an intravenous infusion on a standard dose and schedule (weekly, with the first dose at 400 mg/m2 and all subsequent weekly doses at 250 mg/m2). Dasatinib will be administered orally on a continuous schedule at the following dose levels: 100 mg QD (once a day), 150 mg QD, and 200 mg QD. Three to six patients will be enrolled at each dose level, and the final recommended phase II cohort will be expanded to include up to 12 additional patients. The doses will be escalated in successive cohorts of patients. On cycle 1, dasatinib administration will start one day prior to cetuximab administration. One cycle will be defined as 21 days, and cycles will continue until progression of disease or intolerable toxicities occur. Peripheral blood samples and pharmacokinetic blood samples will be taken on days 0, 1, 15, and 16 of Cycle 1 only. In patients with accessible tumor that give consent, patients will undergo a baseline tumor biopsy and a repeat biopsy after 14-21 days of the first cycle.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed solid malignancy which is recurrent or metastatic or resistant to therapy. Patients w/plan of surgery for recurrent disease post cetuximab/dasatinib are eligible providing that they receive at least 2 cycles of therapy and provide baseline and post-treatment tumor tissue for correlatives.
2. Any number of prior regimens but no prior EGFR or src inhibitors.
3. Age greater or equal to 18 years.
4. ECOG performance status less than or equal to 2 (Karnofsky greater than or equal to 60%).
5. Life expectancy greater than 12 weeks.
6. Patients must have normal organ and marrow function:

   * leukocytes greater than or equal to 3,000/mcL
   * absolute neutrophil count greater than or equal to 1,500/mcL
   * platelets greater than or equal to 100,000/mcL
   * total bilirubin within normal institutional limits
   * AST(SGOT)/ALT(SGPT) less than or equal to 2.5 X institutional upper limit of normal
   * creatinine up to 1.5 x normal institutional limits
7. Ability to understand and the willingness to sign a written informed Consent document.
8. No concomitant medication that are CYP3A4 inducers or potent inhibitors and should not take proton pump inhibitors and H2 antagonists in the first cycle of therapy and should try to avoid taking proton pump inhibitors and H2 antagonists during rest of treatment period.
9. Sexually active women of childbearing potential must use an effective method of birth control during the course of the study, in a manner such that risk of failure is minimized. All WOCBP must have a negative pregnancy test prior to first receiving investigational product.

Exclusion Criteria:

1. Chemotherapy or radiotherapy within 3 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
2. Any other concurrent investigational agents.
3. Patients w/ untreated brain metastases. However, patients who have stable brain disease (should be off corticosteroids) at least 4 weeks after completion of appropriate therapy are eligible.
4. History of allergic reaction to monoclonal antibodies.
5. Inability to swallow oral medications unless patients use a feeding tube.
6. Uncontrolled angina or hypertension or any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or Torsades de pointes).
7. Prolonged QTc interval on pre-entry electrocardiogram (greater than 450 msec) on both the Fridericia and Bazett's correction.
8. Diagnosed or suspected congenital long QT syndrome.
9. Patients currently taking drugs that are generally accepted to have a risk of causing Torsades de Pointes including: quinidine, procainamide, disopyramide, amiodarone, sotalol, ibutilide, dofetilide, erythromycins, clarithromycin, chlorpromazine, haloperidol, mesoridazine, thioridazine, pimozide, cisapride, bepridil, droperidol, methadone, arsenic, chloroquine, domperidone, halofantrine, levomethadyl, pentamidine, sparfloxacin, lidoflazine.
10. Any other uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, or psychiatric illness/social situations that would limit compliance with study requirements.
11. History of significant bleeding disorder unrelated to cancer, including: diagnosed congenital bleeding disorders (e.g., von Willebrand's disease), diagnosed acquired bleeding disorder within one year (e.g., acquired anti-factor VIII antibodies).
12. HIV-positive patients receiving combination antiretroviral therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2007-06; Primary Completion 2009-07 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
To determine the toxicities and the maximum tolerated doses of dasatinib when combined with cetuximab for the treatment of advanced solid tumors | Anticipated completion date December 2008

SECONDARY OUTCOMES:
To determine the objective response rate and overall survival in patients enrolled in the study | Anticipated completion date December 2008
To evaluate tissue biomarkers that relate to EGFR and Src signaling pathways on baseline tumor tissue and to study their modulation with cetuximab/dasatinib on post-treatment tumor tissue | Anticipated completion date December 2008
To measure Src in peripheral blood mononuclear cells (PBMCs) before and after therapy | Anticipated completion date December 2008
To evaluate EGFR gene copy number by FISH on baseline tumor tissue | Anticipated completion date December 2008
To determine pharmacokinetic parameters of dasatinib in patients with and without feeding tubes | Anticipated completion date December 2008

CONTACTS AND LOCATIONS:
Overall Officials: Edward Chu, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Cancer Institute - Hillman Cancer Center, Pittsburgh, Pennsylvania, United States